CLINICAL TRIAL: NCT01048372
Title: An Observational Study to Determine the In-vitro Immunologic and Virology Activity of Cytolin
Brief Title: Observational Study of Blood Treated With Cytolin
Status: Completed | Type: Observational
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009-P-0023471
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: HIV; monoclonal antibody; immune therapy; pathogenesis; cytotoxic T lymphocyte; anti-CD4; anti-self; viral replication; Acute Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early HIV infection: HIV infected adults with early evidence of suppressed cell-mediated immunity but whose disease has not progressed far enough to indicate antiretroviral therapy.
- Control: Healthy adults without HIV infection.

SUMMARY:
Primary Objective: To determine the mechanism of Cytolin's effect on HIV replication from blood drawn from HIV-positive and HIV-negative individuals after exposure to Cytolin.

DETAILED DESCRIPTION:
The initial phase of this in vitro study regarding the potential mechanisms of action of Cytolin was completed in January 2011. Given the data set to date, a decision has been made to extend the study. The extension will allow the Company to further confirm and extend the initial findings regarding the potential mechanism of action of Cytolin.

ELIGIBILITY:
Early HIV Infection

Inclusion Criteria:

* HIV seropositive
* viral load < 100,000 copies/ml
* CD4+ > 350 cells/ul
* Ability and willingness to give written informed consent.

Control Group

Inclusion Criteria:

* HIV seronegative subjects identified as HIV uninfected by a nonreactive HIV 1/2 ELISA.
* Ability and willingness to give written informed consent.

Exclusion Criteria:

* Presentation with an opportunistic infection or AIDS-defining illness.
* Receipt of investigational research agent within 30 days prior to study entry.
* Prior receipt of experimental HIV vaccine, sham vector or adjuvant.
* Receipt of immunosuppressive medications or immune modulators within the past six months. Individuals taking corticosteroid nasal spray for allergic rhinitis, topical steroid or over the counter medications for acute, uncomplicated dermatitis for a period no longer than 14 days will not be excluded.
* Active drug or alcohol use, dependence or psychiatric illness that in the opinion of the study investigator would interfere with adherence to study protocol.
* Serious illness requiring hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult human subjects willing and able to have blood drawn at Massachusetts General Hospital in Boston, MA at baseline, three months and six months. All healthy volunteers have been enrolled and enrollment is now open only to subjects with earlyh HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
T cell number and effector functions in Cytolin-treated blood harvested from HIV infected individuals. | Entry, 3 months, 6 months

SECONDARY OUTCOMES:
In-vitro suppression of viral replication following Cytolin treatment of blood harvested from HIV infected individuals. | Entry, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Rosenberg, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Zarling JM, Ledbetter JA, Sias J, Fultz P, Eichberg J, Gjerset G, Moran PA. HIV-infected humans, but not chimpanzees, have circulating cytotoxic T lymphocytes that lyse uninfected CD4+ cells. J Immunol. 1990 Apr 15;144(8):2992-8. PMID 1969880
- [Background] Morimoto C, Rudd CE, Letvin NL, Schlossman SF. A novel epitope of the LFA-1 antigen which can distinguish killer effector and suppressor cells in human CD8 cells. Nature. 1987 Dec 3-9;330(6147):479-82. doi: 10.1038/330479a0. PMID 2446140
- [Background] Cavallin F, Traldi A, Zambello R. Phenotypical and functional evaluation of CD8+/S6F1+ T lymphocytes in haemophiliac individuals with HIV-1 infection. Clin Exp Immunol. 1993 Jul;93(1):51-5. doi: 10.1111/j.1365-2249.1993.tb06496.x. PMID 8324903
- [Background] Tsubota H, Lord CI, Watkins DI, Morimoto C, Letvin NL. A cytotoxic T lymphocyte inhibits acquired immunodeficiency syndrome virus replication in peripheral blood lymphocytes. J Exp Med. 1989 Apr 1;169(4):1421-34. doi: 10.1084/jem.169.4.1421. PMID 2784486
- [Background] Allen AD, Hart DN, Hechinger MK, Slattery MJ, Chesson CV 2nd, Vidikan P. Leukocyte adhesion molecules as a cofactor in AIDS: basic science and pilot study. Med Hypotheses. 1995 Aug;45(2):164-8. doi: 10.1016/0306-9877(95)90065-9. PMID 8531839
- [Background] Allen AD, Hillis T, Vidikan P, Beer V. Pitfalls in the use of surrogate markers for human immunodeficiency virus disease: further evidence on pathogenesis. Med Hypotheses. 1996 Jul;47(1):27-30. doi: 10.1016/s0306-9877(96)90038-9. PMID 8819112